CLINICAL TRIAL: NCT03594838
Title: Feasibility, Acceptability, Effectiveness and Cost-analysis of Models of HCV Viremia Testing for Confirmation and Cure Among People Who Inject Drugs (PWID): the HEAD*-Start Trial in Georgia
Brief Title: Evaluation of HCV Viremia Testing Approaches Among PWID in Georgia
Acronym: HEAD-Start
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Collaborators: The National Center for Disease Control and Public Health (Unknown); Health Research Union (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 8157-3/1
Record Dates: First submitted 2018-06-13; First posted 2018-07-20 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Hepatitis C, Chronic
Keywords: HCV viremia testing
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Intervention Model Description: A non-randomized 3 arm-interventional study at eight HRSs to evaluate two novel approaches of HCV viremia testing and compare them to the current standard of care. The HRS will be assigned to one of three study arms.
  Six HRSs will provide HCV viremia testing on-site using one of two approaches as follows and two HRS will refer patients off-site for testing (current standard of care).
  The three arms will be compared to determine differences in the proportion of anti-HCV-positive patients that receive HCV viremia test results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Decentralized testing approach (Experimental): Harm reduction site HCV viremia testing approach A. Four HRS will conduct blood draw and point-of-service (decentralized) HCV RNA testing, and results will be provided at the HRS on the same or the following day.
  Interventions: Other: HCV viremia testing approaches
- Centralized testing approach (Experimental): Harm reduction site HCV viremia testing approach B. Two sites will collect blood samples on site and transport them to a reference (centralized) laboratory for HCV viremia testing. Results will be provided at a follow-up visit to the HRS as soon as results are available.
  Interventions: Other: HCV viremia testing approaches
- Standard of Care (No Intervention): Current standard of care. Patients who screen anti-HCV positive at HRS will be referred to HCV treatment centers for HCV RNA testing, and results will be provided at a follow-up visit to the treatment center.

INTERVENTIONS:
Other: HCV viremia testing approaches — Blood draw and HCV viremia testing is done at point of service (Intervention A) Blood draw at point of service and HCV viremia testing at a centralized laboratory (Intervention B)
  Arms: Centralized testing approach; Decentralized testing approach

SUMMARY:
This study will evaluate two novel approaches to improve access to Hepatitis C virus (HCV) confirmatory viremia testing. Both approaches are "Harm reduction site-based (HRS)" because HCV viremia testing will be initiated and test results will be provided at the HRSs. These approaches will be compared to the current standard of care (control) in which anti-HCV-positive individuals must travel to a HCV treatment centre for HCV viremia testing. The investigators hypothesize that improving access to viremia testing improves linkage to care and reduces loss to follow-up among those who screen anti-HCV-positive.

DETAILED DESCRIPTION:
A major step in identifying HCV infected individuals in Georgia has already been implemented by providing rapid anti-HCV testing for people who inject drugs (PWID) at HRS. However, access to HCV confirmatory viremia testing remains limited as PWID must be referred to treatment centers for testing.

Two novel approaches to improve access to HCV viremia testing will be evaluated.

In the first approach, participants with a positive anti-HCV test will have blood drawn and HCV RNA test performed at the HRS. Test results will be provided the same day (or the following day if the participant is unable to wait for results) at the HRS.

In the second approach participants with a positive anti-HCV test will have blood drawn at the HRS. The blood will be processed on site and a plasma sample shipped to a central laboratory for viremia testing. Test results will be communicated to the participants by HRS staff at a follow-up visit as soon as the results are available.

In both groups, participants who test positive will be referred to a treatment centre for further assessments and subsequent treatment initiation.

ELIGIBILITY:
1. People who inject drugs attending for care and needle provision at harm reduction sites.

   Inclusion criteria:
   * Any history of injection drug use (IDU)
   * Age ≥18 years
   * Anti-HCV-positive on rapid diagnostic test performed at the HRS
   * Eligible for the Georgia HCV State Program
   * Living in the catchment area served by the HRS
   * No plans to move out of the catchment area during the next 6 months
   * Willing and able to give informed consent

   Exclusion criteria:
   * Tested HCV RNA-positive from April 2015
   * Pregnancy (self-report)
   * Currently on treatment for hepatitis C
   * Unable to provide a blood sample
2. HRS staff involved in HCV testing and care:

   Inclusion criteria
   * Provide HCV services at HRS from screening through linkage to care.
3. Laboratory staff performing HCV viremia testing at the HRSs, Lugar Centre and Treatment centres:

Inclusion criteria:

* Perform HCV viremia testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1672 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-07-21 (Actual)

PRIMARY OUTCOMES:
HCV care cascade | 6 months
  1.1. Proportion of participants with a positive HCV viremia test who complete each subsequent step in the HCV care cascade
HCV confirmatory viremia test result receipt | 1-30 days
  Proven superiority (with a margin of 10%) of the proportion of participants with a positive anti-HCV test who receive results of an HCV confirmation of viremia test in each intervention arm separately, compared to referral-based testing (SOC)

SECONDARY OUTCOMES:
Entry into HCV care | 1-14 days
  Proven superiority (with a margin of 10%) of the proportion of participants with positive anti-HCV test who submit a blood sample for viremia testing in each intervention arm separately, compared to referral based testing (SOC)
Treatment Initiation Fraction | 4 weeks
  Proportion of participants with positive HCV viremia test who initiate hepatitis treatment
HCV confirmatory viremia test result receipt by intervention | 1-14 day
  Proportion of participants with a positive anti-HCV test who receive results of an HCV confirmation of viremia test using decentralized HCV RNA testing compared to centralized HCV core antigen
Cost of HCV confirmatory viremia testing approach | 6 months
  Costs of HCV viremia testing approaches from a health service and patient perspective
Operational performance of HCV confirmatory viremia testing | 6 months
  Testing volumes at the harm reduction sites
Uptake of HCV confirmatory viremia testing | 4-8 weeks
  Facilitators and barriers of getting an HCV confirmatory viremia test as perceived by participants and health care workers
Attitudes and preferences of participants for HCV confirmatory viremia testing as assessed on a Likert scale | 4-8 weeks
  Willingness of participants to get HCV confirmatory viremia testing as assessed on the Likert Scale of 'strongly agree' (0), 'agree' (1), 'neither agree nor disagree' (2), 'disagree' (3), 'strongly disagree' (4)

CONTACTS AND LOCATIONS:
Overall Officials: Sonjelle Shilton, Study Director — Find; Irma Khonelidze, Principal Investigator — National Centre for Disease Control, Georgia
Locations (8):
- Georgia (8):
  - Imedi Harm Reduction Site, Batumi
  - Step to the Future Harm Reduction Site, Gori
  - New Way Harm Reduction Site, Kutaisi
  - New Vector Harm Reduction Site, Rustavi
  - Akeso Harm Reduction Site, Tbilisi
  - New Vector Harm Reduction Site, Tbilisi
  - New Way Harm Reduction Site, Tbilisi
  - Xenon Harm Reduction Site, Zugdidi